CLINICAL TRIAL: NCT05778630
Title: Emotions and Cognitions in Pediatric Chronic Physical Conditions - the Creation and Implementation of a Psychological Intervention
Brief Title: Emotions and Cognitions in Pediatric Chronic Physical Conditions
Acronym: EmCog
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/14JUI/269; 813546 (Other Grant/Funding Number: European Union Horizon 2020 Program)
Record Dates: First submitted 2021-09-21; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Multiple Chronic Conditions
Keywords: pediatric; chronic disease; intervention; emotion; cognition
MeSH Terms: conditions — Multiple Chronic Conditions; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Individual qualitative interviews. Focus group meetings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A. Focus group (Other): Individuals will participate in one or several, semi-structured focus group meetings.
  Interventions: Other: Focus group meetings; Other: Individual interviews
- Group B. Individual (Other): Individuals will participate in a semi-structured qualitative interview.
  Interventions: Other: Focus group meetings; Other: Individual interviews

INTERVENTIONS:
Other: Focus group meetings — Focus group meetings with different experts in the domain of CPCs (health care professionals) and/or parents or family members of a child with CPC. Focus group meetings will be facilitated by one or two study investigators. Group discussions will be audio-recorded.
Other: Individual interviews — Individual qualitative interviews (semi-directive), conducted by one or two study facilitators.

SUMMARY:
Children living with a chronic physical condition (CPC) are more likely than their peers without a disease to develop psychological difficulties or disorders (Hysing et al., 2007). To prevent or treat these difficulties and disorders, many psychotherapeutic approaches have been developed and tested. Most of them follow a categorical approach, based on a global diagnosis (e.g., Moreira et al., 2013). Few interventions are conducted from a processual perspective (Nef et al., 2012) studying underlying mechanisms of psychological functioning. Emotions and cognitions represent such underlying processes and play an important role in many psychopathological disorders. These processes can weaken but also protect a child from developing psychological difficulties, depending on whether they are effective or not (Gipson et al., 2006; Hysing et al., 2007; Lahaye et al., 2011). The present research project aims to identify a psychological intervention that builds on knowledge of emotional and cognitive processes, considered as protective and risk factors, to prevent/treat psychological difficulties. The project will be conducted in two parts:

1. The first phase aims to better understand the action mechanisms of psychological interventions, focused on emotional and cognitive difficulties of children with CPCs. First, a systematic review will identify recent literature which reports the efficacy of psychological interventions which focused on emotional and cognitive processes. Second, interviews with experts (e.g., pediatricians, psychiatrists, psychologists, nurses, educators) in the field of CPCs and with parents/families of children with CPCs will be conducted. Individual and focus group meetings will be organized, with the aim of identifying the needs of children, based on clinical and practical knowledge and experience. A third phase will consist of the selection of an intervention that will be based on the results of the first two phases.
2. In the second part (not yet registered), the selected intervention will be set up for a feasibility study (Bowen et al., 2009). For this, a small sample of children will participate in the intervention. Participants will be randomly allocated to an intervention group and a control group. The control group will participate in an alternative intervention (e.g., information on chronic diseases). The exact content of the intervention and its form (number of sessions, duration etc.) will be determined by the focus group. The intervention's efficacy will be evaluated (evaluation of emotional and cognitive processes as well as psychological and physiological health), using a mixed method approach. The results will be analyzed and discussed with the focus group. Limitations and perspectives will be formulated to allow for possible transfer of the intervention for future use or to other areas of psychology (Durlak & DuPre, 2008).

DETAILED DESCRIPTION:
The research project will be conducted as a non-medical intervention study, based on a mixed method and action-research principles (Bradbury & Lifvergren, 2016; Ivankova & Wingo, 2018; Malengreaux et al., 2020; Marshall et al., 2006). It will include a systematic literature review, quantitative (standardized questionnaires, self and hetero-reports) and qualitative measures (dialogues and discussions, semi-directed interviews, audio-recordings, observations, written reports). The effectiveness study of PART II of the research project will be carried out as randomized controlled trial but is not described in this registration.

PART 1

Phase I.a:

A systematic literature review is conducted by all investigators (researchers) in order to better understand action mechanisms of psychological interventions for children with chronic diseases (registered in PROSPERO: CRD42021233505).

Phase I.b:

* Individual semi-structured qualitative interviews will be conducted by one or two investigators to explore the following questions: Which are emotional and cognitive difficulties and resources in children with CPC? Which are the emotional and cognitive needs of children with CPC? How are these/can these be addressed?
* One or several focus groups will be created. They will be composed of different experts in the domain of CPCs (health care professionals, families, researchers, etc.). Per group, one or several meetings will be organized, depending on participants' availabilities. The meetings will be conducted by one or two investigators who will use semi-structured interview techniques to explore the following questions: Which are emotional and cognitive difficulties and resources in children with CPC? Which are the emotional and cognitive needs of children with CPC? How are these/can these be addressed?

PART II will consist of a feasibility and an effectiveness study of the intervention. For both studies, the selected intervention will be implemented, based on scientific, rigorous methods, and be evaluated with different quantitative and qualitative measures. PART II will rely on PART I. Thus, it will be described in another registration after completion of PART I.

ELIGIBILITY:
Inclusion criteria:

The participant

* is a health care professional in the domain of pediatric chronic diseases or parents/family members/tutors of a child with CPC, aged 8-12 years OR
* is in regular contact with children with a chronic physical condition who are between 8 and 12-years-old.
* speak fluently French

Exclusion Criteria:

* Health care professionals who are not in regular contact with children, 8 to 12 years- old, with a chronic physical condition
* Parents with a child with CPC who is not 8 to 12 years old
* Participants who do not speak French

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Interview data outcomes | October 2021-December 2024
  Interview questions will explore: 1) emotional and cognitive difficulties and resources of children with CPC, 2) emotional and cognitive needs of children with CPC. Audio data from semi-structured group meetings and semi-structured individual interviews will be transcribed and analysed with thematic analysis (Braun & Clarke, 2006).

SECONDARY OUTCOMES:
Interview data outcomes and systematic review results | October 2021-December 2024
  Narrative comparison of emerged themes from the thematic analysis of qualitative interview data, to results of the systematic literature review.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Moniotte, Principal Investigator — Cliniques universitaires Saint-Luc UCLouvain
Locations (1):
- Mareike Kaemmerer, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sansom-Daly UM, Peate M, Wakefield CE, Bryant RA, Cohn RJ. A systematic review of psychological interventions for adolescents and young adults living with chronic illness. Health Psychol. 2012 May;31(3):380-93. doi: 10.1037/a0025977. Epub 2011 Nov 7. PMID 22059621
- [Background] McNally K, Rohan J, Pendley JS, Delamater A, Drotar D. Executive functioning, treatment adherence, and glycemic control in children with type 1 diabetes. Diabetes Care. 2010 Jun;33(6):1159-62. doi: 10.2337/dc09-2116. Epub 2010 Mar 9. PMID 20215458
- [Background] Marshall, P., de Salas, K., & Mckay, J. (2006). Action research in practice: Balancing the dual imperatives. ACIS 2006 Proceedings - 17th Australasian Conference on Information Systems.
- [Background] Lahaye M, Van Broeck N, Bodart E, Luminet O. Predicting quality of life in pediatric asthma: the role of emotional competence and personality. Qual Life Res. 2013 May;22(4):907-16. doi: 10.1007/s11136-012-0194-7. Epub 2012 May 15. PMID 22585190
- [Background] Luminet, O. (2008). Psychologie des émotions (2nd edition). De Boeck.
- [Background] Nef, F., Phillippot, P., & Verhofstadt, L. (2012). L'approche processuelle en évaluation et intervention cliniques: une approche psychologique intégrée. Revue Francophone de CliniqueComportementale et Cognitive, 17(3). http://hdl.handle.net/2078.1/129174
- [Background] Thabrew H, Stasiak K, Hetrick SE, Donkin L, Huss JH, Highlander A, Wong S, Merry SN. Psychological therapies for anxiety and depression in children and adolescents with long-term physical conditions. Cochrane Database Syst Rev. 2018 Dec 22;12(12):CD012488. doi: 10.1002/14651858.CD012488.pub2. PMID 30578633
- [Background] Beale IL. Scholarly literature review: Efficacy of psychological interventions for pediatric chronic illnesses. J Pediatr Psychol. 2006 Jun;31(5):437-51. doi: 10.1093/jpepsy/jsj079. Epub 2005 Sep 14. PMID 16162841
- [Background] Plante WA, Lobato D, Engel R. Review of group interventions for pediatric chronic conditions. J Pediatr Psychol. 2001 Oct-Nov;26(7):435-53. doi: 10.1093/jpepsy/26.7.435. PMID 11553698
- [Background] Hysing M, Elgen I, Gillberg C, Lie SA, Lundervold AJ. Chronic physical illness and mental health in children. Results from a large-scale population study. J Child Psychol Psychiatry. 2007 Aug;48(8):785-92. doi: 10.1111/j.1469-7610.2007.01755.x. PMID 17683450
- [Background] Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative Research in Psychology, 3(2), 77-101. https://doi.org/10.1191/1478088706qp063oa